# Non-Interventional Study

### A5481188

Impact of age and comorbidities on treatment outcomes of first-line treatment with palbociclib in combination with an aromatase inhibitor (AI) in patients diagnosed with HR+/HER2 - metastatic breast cancer – Danish Non-Interventional Study

# Statistical Analysis Plan

(SAP)

Version: 1.0

Author: PPD , Pfizer Denmark

Date: 1-Mar-2024

## **TABLE OF CONTENTS**

| 1. LIST OF ABBREVIATIONS | 3 |
|-------------------------------------------|----|
| 2. RATIONALE AND BACKGROUND | 4 |
| 3. STUDY OBJECTIVES AND HYPOTHESES | 4 |
| 3.1. Primary objectives (all patients) | 4 |
| 3.2. Secondary objectives | 4 |
| 4. RESEARCH METHODS | 5 |
| 4.1. Study design | 5 |
| 4.2. Study population | 5 |
| 4.2.1. Subgroups | 5 |
| 4.3. Variables | 6 |
| 4.4. Data sources | 7 |
| 4.5. Sample size and power calculations | 7 |
| 4.6. Missing Data | 7 |
| 4.7. Statistical methodology and analyses | 7 |
| 4.7.1. Index date and follow-up | 7 |
| 4.7.2. Primary analyses | 8 |
| 4.7.3. Secondary analyses | 8 |
| 4.7.4. Post-hoc analyses | 10 |
| 5. REFERENCES | 10 |
| 6. APPENDICES | 11 |
| 6.1. Appendix A: Table shells | 11 |
| 6.2 Appendix B: Additional information | 15 |

## 1. LIST OF ABBREVIATIONS

| Abbreviation | Definition |
|---|---|
| AI | Aromatase Inhibitor |
| CCI | Charlson Comorbidity Index |
| CDK4 | Cyclin Dependent Kinase 4 |
| CDK6 | Cyclin Dependent Kinase 6 |
| CI | Confidence interval |
| DBCG | Danish Breast Cancer Group |
| DC50 | ICD-10 code for patients with breast cancer |
| EC | European Commission |
| EMA | European Medicines Agency |
| HR | Hormone receptor; hazard ratio |
| HR+ | Hormone receptor positive, including estrogen receptor positive (ER+) |
| HER2 | Human epidermal growth factor receptor 2 |
| HER2- | HER2 negative |
| LOT | Line of Treatment |
| mBC | Metastatic breast cancer |
| NIS | Non-Interventional Study |
| OS | Overall survival |
| PFS | Progression free survival |
| RCT | randomized controlled trials |
| RW | Real-World |
| RWE | Real-World Evidence |

### 2. RATIONALE AND BACKGROUND

Strict inclusion and exclusion criteria in clinical trials restricts inclusion of elderly patients as well as patients with certain comorbidities. With this there is an unmet need. The impact of comorbidities on palbociclib effectiveness has recently been studied in a number of real-world observational studies from the US.

In a Danish setting, limited evidence is available on older metastatic breast cancer patients with comorbidities and the effectiveness of treatment with palbociclib in these subgroups of the Danish mBC patients. As an update and extension of the Garly et al. study (3), the present study therefore aims to investigate the use and effectiveness of palbociclib in all HR+/HER2- mBC patients in Denmark, as well as in subgroups of elderly patients and those with comorbidities. The study data will be based on the DBCG clinical database as the previous study by Garly et al. (3).

### 3. STUDY OBJECTIVES AND HYPOTHESES

Utilizing the DBCG register the overall objective is to retrospectively investigate the outcomes (overall PFS and OS) of first-line treatment with palbociclib in combination with an aromatase inhibitor (AI) in key subgroups of mBC patients in Denmark focusing on age and comorbidity burden.

## 3.1. Primary objectives (all patients)

- PFS of all mBC patients receiving palbociclib in combination with AI as first-line treatment
- OS of all mBC patients receiving palbociclib in combination with AI as first-line treatment

## 3.2. Secondary objectives

- Age subgroup analyses:
  - Age distribution in the full data set of mBC patients receiving palbociclib + AI as firstline treatment
  - PFS and OS in mBC patients below 65 years of age, 65-74 years of age and 75+ years of age, respectively, receiving palbociclib + AI as first-line treatment
- Comorbidity subgroup analyses (Charlson Comorbidity Index (CCI) (4) is used as a data source for comorbidity and comorbidity burden – comorbidities at the start of palbociclib treatment):
  - PFS and OS in the full data set of mBC patients receiving palbociclib + AI as first-line treatment split into Charlson Comorbidity Index (CCI) point scores of 0, 1, 2, and 3 or higher (3+)
  - PFS and OS in the full data set of mBC patients receiving palbociclib + AI as first-line treatment split into number of comorbidities (no comorbidity, one comorbidity, and two or more comorbidities)
  - PFS and OS in the full data set of mBC patients receiving palbociclib + AI as first-line treatment split into type of comorbidity – focus on five main groups: Cardiac disease, Vascular disease, Metabolic disease, Psychiatric disease, Blood and lymphatic system.

### 4. RESEARCH METHODS

## 4.1. Study design

The study is designed as a secondary data collection non-interventional study (NIS). Retrospective data will be collected from an existing registry - the Danish Breast Cancer Group (DBCG) registry. The focus of this study will be on HR+/HER2- locally advanced or metastatic breast cancer treated with palbociclib. The study is a single-arm study focusing on patients treated with palbociclib in Denmark.

## 4.2. Study population

In the DBCG registry, all HR+/HER2- locally advanced or mBC patients treated with palbociclib in combination with AI as first-line treatment will be identified. Palbociclib was approved by the European Commission (EC) and European Medicines Agency (EMA) in November 2016. Hence, the study period will be from 1 January 2017 and to 31 December 2021. A follow-up on patients until 31 December 2023 in terms of the estimation of PFS and OS will be made. The study will only include patients treated with palbociclib+AI as first-line treatment.

#### Inclusion Criteria

Patients must meet the following inclusion criteria to be eligible for inclusion in the study:

- Patients with breast cancer (ICD-10: DC50)
- A diagnosis of HR+/HER2- locally advanced or metastatic breast cancer
- 3. Endocrine sensitive, endocrine resistant, or de novo mBC patient
- Initiated treatment with palbociclib as first-line treatment (palbociclib + AI) between 1
  January 2017 and 31 December 2021
- Inclusion data: Data of relapse/stage IV disease/progression leading to initiation of palbociclib+AI

#### Exclusion Criteria

There are no exclusion criteria for this study.

### 4.2.1. Subgroups

Besides presenting results for all mBC patients treated with palbociclib in combination with Al patients as first-line treatment results for different subgroups split by age and comorbidities as well as disease-specific characteristics will also be presented.

These subgroups of HR+/ HER2 negative mBC patients are:

- Patients below 65 years of age
- Patients 65-74 years of age
- Patients 75+ years of age
- Patients split by comorbidity severity score (CCI; 0, 1, 2, and 3 or higher (3+))
- Patients split by number of comorbidities (0, 1, 2+)
- Patients split in types of comorbidities (Cardiac disease, Vascular disease, Metabolic disease, Psychiatric disease, Blood and lymphatic system)
- Patients with or without visceral disease
- Bone only patients
- Endocrine resistant, endocrine sensitive or de novo patients

## 4.3. Variables

The main variables included in the study are the following:

| Variable | Role | Data source(s) | DBCG<br>variable(s) |
|---|---|---|---|
| Diagnosis (ICD-10 code: DC50) | Exposure/<br>Inclusion | DBCG registry | Not applicable |
| Treatment with palbociclib | Exposure/<br>Inclusion | DBCG registry | RE201, RE201A |
| Date of birth | Baseline | DBCG registry | Based on M1 |
| Date of breast cancer diagnosis | Baseline | DBCG registry | Not applicable |
| Occurrence of metastases | Baseline | DBCG registry | RE220-RE227 |
| Visceral status (visceral and non-visceral – visceral defined as metastases in the organs, e.g., lung, liver)) | Baseline | DBCG registry | RE220-RE227 |
| Bone only | Baseline | DBCG registry | RE14 |
| Metastatic sites (liver, lung, CNS, lymph nodes) | Baseline | DBCG registry | RE10-18 + 80-81,<br>117-119, 219-222 |
| Endocrine resistant (recurrent pts with advanced disease within 12 months of completing adjuvant endocrine therapy) | Baseline | DBCG registry | Calculated |
| Endocrine sensitive (recurrent pts with advanced disease after 12 months of completing adjuvant endocrine therapy, recurrent pts who received no adjuvant endocrine therapy) | Baseline | DBCG registry | Calculated |
| De Novo (primary mBC – newly metastatic) | Baseline | DBCG registry | Calculated |
| Date of relapse | Baseline | DBCG registry | RE1-RE3 |
| Date for treatment initiation with palbociclib | Baseline | DBCG registry | RE203-RE205 |
| Date for treatment stop with palbociclib | Baseline | DBCG registry | RE206-RE208 |
| Charlson Comorbidity Index (CCI) – point scores of 0, 1, 2 and 3 or higher (3+) (calculated at start of palbociclib treatment) | Baseline | National Patient Registry<br>data used to define CCI<br>in DBCG registry | Not applicable |
| Number of comorbidities (calculated at start of palbociclib treatment) | Baseline | National Patient Registry<br>data used to define CCI<br>in DBCG registry | Not applicable |
| Types of comorbidities (Cardiac disease, Vascular disease, Metabolic disease, Psychiatric disease, Blood and lymphatic system) (at start of palbociclib treatment) | Baseline | National Patient Registry<br>data used to define CCI<br>in DBCG registry | Not applicable |
| Death date | Baseline<br>charac. | DBCG registry | Not applicable |
| PFS (see section 8.1 for definition) | Outcome | Estimated via DBCG registry | Based on<br>variables listed in<br>this table |
| OS (see section 8.1 for definition) | Outcome | Estimated via DBCG registry registrations | Based on<br>variables listed in<br>this table |

### 4.4. Data sources

This study will be based on the DBCG clinical database and the National Patient Registry (LPR) with respect to the comorbidities. Data from the DBCG clinical database and the National Patient Registry will be combined by the personal identification codes (CPR)) that every Danish citizen has.

## 4.5. Sample size and power calculations

The study is purely descriptive and explorative. No formal hypotheses will be tested in the study. Calculation of sample size is therefore not applicable.

The expected and estimated total study population with the focus on all Danish mBC patients (endocrine sensitive, endocrine resistant or de novo) that have received palbociclib in combination with AI as first-line therapy. 580 patients will be included from 1 January 2017 to 31 December 2021.

Subgroup analyses of this patient population will be made based on age and comorbidity.

## 4.6. Missing Data

The study will only include patients for whom there are complete registrations in the DBCG register. However, should missing data occur, no imputation will be made, and all statistics will be calculated with non-missing values. Counts and percentages of missing values will be presented in the tables where applicable.

### 4.7. Statistical methodology and analyses

The study is a single-arm study and will be purely descriptive and explorative. No formal hypotheses will be tested.

This study will provide two types of outcomes:

- Outcomes on PFS and OS of patients treated with palbociclib+Al as first-line (population and subpopulations (Age and Comorbidity) (Appendix A, Table 3 and 4))
- Descriptive statistics on the population/subpopulations treated with palbociclib+Al (Appendix A, Table 1 and 2)

## 4.7.1. Index date and follow-up

Definitions of the incidence data and the index date of the first-line treated palbociclib + Al patients shown together with the definition of the treatment outcomes (PFS and OS), as well as definition of visceral disease can be found in the table below.

| Incidence date | The date of the initial breast cancer diagnosis. |
|---|---|
| Index date | The date of relapse or stage IV disease. |
| Progression Free<br>Survival (PFS) | The time from the date of relapse or stage IV disease (index date) to progression or death, whichever occurs first. Patients will be censored 31 December 2021. Progression is based on radiological, clinical, and biochemical examination from the treating departments. |
| Overall Survival (OS) | The time from index date to death at any cause. |
| Visceral disease | Defined as metastases in the organs, e.g., lung, liver. Visceral disease is based on the variable Location of metastases (RE10-18 + 80-81, 117-119, 219-222) in the DBCG database. |

For the PFS and OS outcomes for the full palbociclib first-line population (primary analyses) as well as each subpopulation (secondary analyses), as presented below, Kaplan-Meier survival distribution functions with 95% confidence intervals will be estimated. Hence, if possible median PFS and OS as well as interquartile ranges (IQR) will be estimated. Unadjusted Kaplan Meier curves will be presented to illustrate time-to-event (PFS or OS).

For the descriptive statistics, numbers and percentages will be provided and presented in tables, including cross tabulations (see section 6 for presentation of tables shells).

All data analysis will be executed using the statistical software R-studio.

### 4.7.2. Primary analyses

As primary analyses (descriptive) of PFS and OS will be estimated for <u>all</u> Danish mBC patients receiving palbociclib as first-line treatment in combination with AI. PFS will be estimated for all patients until either a physician-assessed disease progression occurred, death or until data cut-off by 31 December 2023. OS will be estimated for all patients with a censoring of data by 31 December 2023 as the last day of data capture in the study.

## 4.7.3. Secondary analyses

Similar to the primary analyses, univariate analyses of PFS and OS for subgroups (age and comorbidity) of all mBC patients having palbociclib + Al as first-line treatment will be made and with the same definitions and timelines for their estimation.

These subgroups of HR+/ HER2 negative mBC patients are:

#### Age-groups

- Patients below 65 years of age
- Patients 65-74 years of age
- Patients 75+ years of age

Statistical test of differences in baseline characteristics as well as the PFS and the OS outcomes between each of these age subgroups compared to all first-line palbociclib patients the Shapiro-Wilk test of normality and the Wilcoxon rank sum will be applied.

Palbociclib
A5481188 NON-INTERVENTIONAL STUDY STATISTICAL ANALYSIS PLAN FOR SECONDARY DATA
COLLECTION STUDY
Version 1.0,1 March 2024

Palbociclib
A5481188 NON-INTERVENTIONAL STUDY STATISTICAL ANALYSIS PLAN FOR SECONDARY DATA
COLLECTION STUDY
Version 1.0,1 March 2024

Comorbidities as measured by Charlson Comorbidity Index (CCI)

- Patients split by comorbidity severity score (CCI; 0, 1, 2, and 3 or higher (3+))
- Patients split by number of comorbidities (0, 1, 2+)
- Patients split in types of comorbidities (Cardiac disease, Vascular disease, Metabolic disease, Psychiatric disease, Blood and lymphatic system)

Statistical test of differences in baseline characteristics as well as the PFS and the OS outcomes between each of these comorbidity groups will be performed, e.g. using the chi-square test).

And finally various disease-specific characteristics of the mBC patients having palbociclib + AI as first-line treatment.

- · Patients with or without visceral disease
- Bone only patients
- Endocrine resistant, endocrine sensitive or de novo patients

Similar statistical test of difference as for the two other subgroups will be made for the disease-specific characteristics.

## 4.7.4. Post-hoc analyses

Not applicable.

### 5. REFERENCES

- Tripathy D, Blum JL, Karuturi MS, McCune S, Kurian S, Moezi MM, Anderson DM, Wang Y, Montelongo MZ, Zhang Z, Gauthier E, Rocque E; Impact of comorbidities on real-world patientreported outcomes of patients with hormone receptor positive human epidermal growth factor 2 negative (HR+/HER2-) advanced breast cancer enrolled in the POLARIS trial. ESMO 2023 373P. https://oncologypro.esmo.org/meeting-resources/esmo-congress/impact-of-comorbidities-on-realworld-rw-clinical-outcomes-of-patients-pts-with-hormone-receptor-positive-human-epidermalgrowth-factor-2-negat.
- Brufsky A, Liu X, Li B, McRoy L, Chen C, Makari D, Layman R, Rugo H; Real-world effectiveness
  of palbociclib plus aromatase inhibitors (AI) in metastatic breast cancer patients with
  cardiovascular diseases. SABCS 2023 PO1-17-05. 2023 SABCS Abstract Report-12-1-23
  (atgproductions.net).
- Garly R, Berg T, Jensen MB, Knoop A, Volmer L, Glavicic V, Khan H, Poulsen PB, Olsen J, Kümler I. A Retrospective, Non-Interventional Study of Breast Cancer Patients Diagnosed With ER+/HER2 Negative, Locally Advanced or Metastatic Breast Cancer Treated with Palbociclib in Denmark. Acta Oncologica 2023;1-8. https://doi:10.1080/0284186X.2023.2194030.
- DMCG.dk Benchmarking Consortium. Rapport om canceroverlevelse i Danmark 1995-2012. https://www.dmcg.dk/siteassets/arsberetninger-og-udgivelser/benchmarking-consortium/a forsider metoder 10 11 2014.pdf

## 6. APPENDICES

# 6.1. Appendix A: Table shells

This section presents an overview of the table shells.

**Table 1.** Descriptive statistics. All mBC patients having palbociclib as first-line treatment in combination with Al

| combination with | | | D# |
|---|---|---|---|
| Population | Subgroup | Outcome | Result |
| All included | All patients | Number of | N (100%) |
| patients | | patients (all) | Madian area and standard |
| (first-line treated with | | Age | Median, mean and standard |
| | | | deviation |
| palbociclib+AI) All included | Patients below 65 years of age | Number of | NI (0/) |
| patients | Patients below 65 years of age | Number of<br>patients | N (%) |
| (first-line treated | Patients 65-74 years of age | Number of | N (%) |
| with | Fallents 65-74 years or age | patients | N (70) |
| palbociclib+AI) | Patients 75+ years of age | Number of | N (%) |
| pariodicino (711) | Fallents 75+ years or age | patients | N (70) |
| All included | Comorbidities 1 | Number of | N (%) in each group |
| patients | - patients split into severity of | patients with | 14 (70) iii each group |
| (first-line treated | comorbidities as measured by | a CCI score | |
| with | CCI (0, 1, 2, 3 or higher (3+)) | of 0, 1, 2, 3 or | |
| palbociclib+AI) | 227 (2, 1, 2, 2 2. 13.1.2. (2 7) | higher (3+), | |
| , | | respectively | |
| | | Age | Median, mean and standard |
| | | " | deviation |
| | Comorbidities 2 | Number of | N (%) in each group |
| | - patients split into number of | patients with | |
| | comorbidities (0, 1, 2+) | 0, 1, or 2+ | |
| | | comorbidities, | |
| | | respectively | |
| | | Age | Median, mean and standard |
| | | | deviation |
| | Comorbidities 3 | Number of | N (%) in each group |
| | - patients split into type of | patients with | N (%) in each group |
| | comorbidities | specific type | |
| | (Cardiac disease, Vascular | of comorbidity | |
| | disease, Metabolic disease, | Age | Median, mean and standard |
| | Psychiatric disease, Blood and | , .gc | deviation |
| | lymphatic system) | | 201122011 |
| All included | Patients with visceral disease | Number of | N (%) |
| patients | | patients | Madian managed at a dead |
| (first-line treated | | Age | Median, mean and standard |
| with | Detients without vices and | Mumber | deviation |
| palbociclib+AI) | Patients without visceral | Number of | N (%) |
| | disease | patients | Madian maan and standard |
| | | Age | Median, mean and standard deviation |
| All included | Datiente hone only | Number of | |
| All included | Patients bone only | | N (%) |
| patients<br>(first-line treated | | patients | Madian mean and standard |
| with | | Age | Median, mean and standard |
| palbociclib+Al) | Endocrino registent nationte | Number of | deviation N (%) |
| paibociciib*Ai) | Endocrine resistant patients | | /V (70) |
| I | | patients | |

| | Age | Median, mean and standard deviation |
|---|---|---|
| Endocrine sensitive patients | Number of<br>patients | N (%) |
| | Age | Median, mean and standard deviation |
| De Novo patients (primary mBC) | Number of<br>patients | N (%) |
| | Age | Median, mean and standard deviation |

**Table 2.** Disease-specific descriptive statistics. All mBC patients having palbociclib as first-line treatment in combination with Al

| Population | Subgroup | Outcome | Result |
|---|---|---|---|
| All included patients | All patients | Type of metastases | Visceral: N (%) |
| (first-line treated with | | | Non-visceral: N (%) |
| palbociclib+AI) | | | Both: N (%) |
| | | Number of metastases | 0: N (%) |
| | | | 1: N (%) |
| | | | 2: N (%) |
| | | | >2: N (%) |
| | | Metastatic site | Skin: N (%) |
| | | | Bone: N (%) |
| | | | Lung: N (%) |
| | | | Liver: N (%) |
| | | | CNS: N (%) |
| | | | Other: N (%) |
| All included patients | Patients below 65 years of age | Type of metastases | Visceral: N (%) |
| (first-line treated with | | | Non-visceral: N (%) |
| palbociclib+Al) | | | Both: N (%) |
| | | Number of metastases | 0: N (%) |
| | | | 1: N (%) |
| | | | 2: N (%) |
| | | | >2: N (%) |
| | | Metastatic site | Skin: N (%) |
| | | | Bone: N (%) |
| | | | Lung: N (%) |
| | | | Liver: N (%) |
| | | | CNS: N (%) |
| | 5 !! | | Other: N (%) |
| | Patients 65-74 years of age | Type of metastases | Visceral: N (%) |
| | | | Non-visceral: N (%) |
| | | Nember | Both: N (%) |
| | | Number of metastases | 0: N (%) |
| | | | 1: N (%) |
| | | | 2: N (%) |
| | | | >2: N (%) |
| | | Metastatic site | Skin: N (%) |
| | | | Bone: N (%) |
| | | | Lung: N (%) |
| | | | Liver: N (%) |
| | | | CNS: N (%) |
| | Patients 75+ years of age | Type of metastases | Other: N (%)<br>Visceral: N (%) |
| | Fauerits 75+ years or age | Type of metastases | Non-visceral: N (%) |
| | | | Both: N (%) |

| | | Number of metastases | 0: N (%) |
|---|---|---|---|
| | | | 1: N (%) |
| | | | 2: N (%) |
| | | 14-4-4-4::4- | >2: N (%) |
| | | Metastatic site | Skin: N (%) |
| | | | Bone: N (%) |
| | | | Lung: N (%) |
| | | | Liver: N (%) |
| | | | CNS: N (%) |
| All included a sticuta | Companidition 4 | Time of metectaria | Other: N (%) |
| All included patients | Comorbidities 1 | Type of metastases | Visceral: N (%) |
| (first-line treated with<br>palbociclib+AI) | - patients split into severity of comorbidities as measured by | | Non-visceral: N (%)<br>Both: N (%) |
| paibociciib+AI) | | l | DUII. N (70) |
| | CCI (0, 1, 2, 3 or higher (3+)) | | |
| | | Number of metastassa | O: N (0/) |
| | | Number of metastases | 0: N (%) |
| | | | 1: N (%) |
| | | | 2: N (%)<br>>2: N (%) |
| | | | ~2. IV (70) |
| | | Metastatic site | Skin: N (%) |
| | | Wetastatic site | Bone: N (%) |
| | | | Lung: N (%) |
| | | | Liver: N (%) |
| | | | CNS: N (%) |
| | | | Other: N (%) |
| | Comorbidities 2 | Type of metastases | Visceral: N (%) |
| | - patients split into number of | Type of metastases | Non-visceral: N (%) |
| | comorbidities (0, 1, 2+) | | Both: N (%) |
| | 55676/did00 (0, 1, 2 · ) | | 2031. 11 (70) |
| | | Number of metastases | 0: N (%) |
| | | | 1: N (%) |
| | | | 2: N (%) |
| | | | >2: N (%) |
| | | Metastatic site | Skin: N (%) |
| | | | Bone: N (%) |
| | | l | Lung: N (%) |
| | | | Liver: N (%) |
| | | | CNS: N (%) |
| | | | Other: N (%) |
| | Comorbidities 3 | Type of metastases | Visceral: N (%) |
| | - patients split into type of | | Non-visceral: N (%) |
| | comorbidities | | Both: N (%) |
| | (Cardiac disease, Vascular disease, | Number of metastases | 0: N (%) |
| 1 | Metabolic disease, Psychiatric<br>disease, Blood and lymphatic | | 1: N (%) |
| I | | I | 2: N (%) |
| | | I | |
| | system) | | >2: N (%) |
| | | Metastatic site | >2: N (%)<br>Skin: N (%) |
| | | Metastatic site | >2: N (%)<br>Skin: N (%)<br>Bone: N (%) |
| | | Metastatic site | >2: N (%)<br>Skin: N (%)<br>Bone: N (%)<br>Lung: N (%) |
| | | Metastatic site | >2: N (%)<br>Skin: N (%)<br>Bone: N (%)<br>Lung: N (%)<br>Liver: N (%) |
| | | Metastatic site | >2: N (%)<br>Skin: N (%)<br>Bone: N (%)<br>Lung: N (%) |

Table 3. Progression Free Survival (PFS)\*. All mBC patients having palbociclib as first-line treatment in combination with Al

| Endpoint | Population | Subgroup | Outcome | Result |
|---|---|---|---|---|
| Primary | All included patients<br>(first-line treated with<br>palbociclib+Al) | All patients | PFS | Median and IQR |
| Secondary | All included patients | Patients below 65 years of age | PFS | Median and IQR |
| | (first-line treated with palbociclib+AI) | Patients 65-74 years of age | PFS | Median and IQR |
| | palbocicilb - / ti/ | Patients aged 75+ years of age | PFS | Median and IQR |
| Secondary | All included patients<br>(first-line treated with<br>palbociclib+Al) | Comorbidities 1 - patients split into severity of comorbidities as measured by CCI (0, 1, 2, 3 or higher (3+)) | PFS | Median and IQR |
| | | Comorbidities 2 - patients split into number of comorbidities (0, 1, 2+) | PFS | Median and IQR |
| | Comorbidities 3 - patients split into type of comorbidities (Cardiac disease, Vascular disease, Metabolic disease, Psychiatric disease, Blood and lymphatic system) | PFS | Median and IQR | |
| Secondary | All included patients (first-line treated with palbociclib+Al) | Patients with visceral disease | PFS | Median and IQR |
| | | Patients without visceral disease | PFS | Median and IQR |
| Secondary | Secondary All included patients (first-line treated with | Patients bone-only | PFS | Median and IQR |
| palbociclib+AI) | Patients not bone-only | PFS | Median and IQR | |
| Secondary All included patients (first-line treated with | Endocrine resistant patients | PFS | Median and IQR | |
| | palbociclib+AI) | Endocrine sensitive patients | PFS | Median and IQR |
| | | De novo patients | PFS | Median and IQR |

Table note: \* Following definition of PFS in section 4.7.1.

**Table 4.** Overall Survival (OS)\*. All mBC patients having palbociclib as first-line treatment in combination with Al

| Endpoint | Population | Subgroup | Outcome | Result |
|---|---|---|---|---|
| Primary | All included patients<br>(first-line treated with<br>palbociclib+Al) | All patients | os | Median and IQR |
| Secondary | All included patients | Patients below 65 years of age | OS | Median and IQR |
| | (first-line treated with palbociclib+AI) | Patients 65-74 years of age | OS | Median and IQR |
| | paisonini 747 | Patients aged 75+ years of age | OS | Median and IQR |
| Secondary All included patients (first-line treated with palbociclib+Al) | Comorbidities 1 - patients split into severity of comorbidities as measured by CCI (0, 1, 2, 3 or higher (3+)) | OS | Median and IQR | |
| | Comorbidities 2 - patients split into number of comorbidities (0, 1, 2+) | os | Median and IQR | |
| | | Comorbidities 3 - patients split into type of comorbidities (Cardiac disease, Vascular disease, Metabolic disease, Psychiatric disease, Blood and lymphatic system) | os | Median and IQR |
| Secondary | All included patients<br>(first-line treated with | Patients with visceral disease | os | Median and IQR |
| | palbociclib+AI) | Patients without visceral disease | OS | Median and IQR |
| Secondary | All included patients | Patients bone-only | OS | Median and IQR |
| | (first-line treated with<br>palbociclib+AI) | Patients not bone-only | os | Median and IQR |
| Secondary | All included patients<br>(first-line treated with<br>palbociclib+Al) | Endocrine resistant patients | os | Median and IQR |
| | | Endocrine sensitive patients | OS | Median and IQR |
| | | De novo patients | OS | Median and IQR |

Table note: \* Following definition of OS in section 4.7.1.

For PFS and OS (Table 3 and 4), unadjusted Kaplan Meier curves will be presented.

## 6.2. Appendix B: Additional information

None.